CLINICAL TRIAL: NCT02950896
Title: Intraoperative Fetal Heart Rate (FHR) Monitoring: a Feasibility Study
Status: Terminated | Type: Observational
Why Stopped: Appropriate devices for fetal heart rate monitoring were not available.
Sponsor: Washington University School of Medicine (Other)
Responsible Party: Sponsor
Other Study IDs: 201606134
Record Dates: First submitted 2016-10-28; First posted 2016-11-01 (Estimated); Results first posted 2019-05-10 (Actual); Last update posted 2019-05-10 (Actual); Status verified 2019-02

CONDITIONS: Fetal Monitoring; Labor, Obstetric

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- intraoperative FHR monitoring: Intraoperative fetal heart rate (FHR) monitoring
  Interventions: Other: observational fetal heart rate monitoring

INTERVENTIONS:
Other: observational fetal heart rate monitoring — Patients will have fetal heart rate monitoring

SUMMARY:
Fetal heart rate [FHR] monitoring is used widely to assess the well-being of the baby in the delivery period. If it is determined that an urgent cesarean delivery is required because of fetal distress, FHR is discontinued once the mother is in the operating room in order to allow for surgical site preparation. From this point, there is no real-time monitoring that permits assessment of the well-being of the infant. The investigators are evaluating the feasibility of intraoperative FHR monitoring using fetal ECG placed on the mother's upper abdominal wall and the standard acoustic device routinely used. The investigators will compare these to the traditional well-being tests: umbilical arterial blood gas and Apgar score.

The first 15 subjects will be recruited from pregnant women who have scheduled induction of labor. The subsequent 40 subjects will be recruited from pregnant women who have scheduled cesarean sections.

DETAILED DESCRIPTION:
Fetal heart rate (FHR) monitoring has become the most widely used assessment of fetal well-being in the peripartum period and the only routinely used method that provides continuous fetal monitoring. Despite a false positive rate for the detection of intrapartum asphyxia leading to cerebral palsy of over 99% [1-3] FHR monitoring continues to be the mainstay of peripartum fetal surveillance. FHR monitoring is routinely available in the operating room, where it is typically reassessed in cases of urgent cesarean delivery for fetal distress since it may direct immediate anesthetic and peripartum management. However, despite the ubiquitous use of FHR monitoring in labor and the typical use of FHR monitoring on arrival to the OR, FHR monitoring is universally stopped once anesthesia has been performed in order to allow abdominal skin preparation and for surgery to proceed. From the moment of anesthesia induction until fetal delivery, no real-time data is available that allows assessment of fetal well-being. A few isolated studies and case reports in the 1970s-1980s examined intraoperative FHR monitoring using scalp-clip electrodes during Cesarean deliveries [4-7]. None of these studies assessed external FHR monitors or current anesthesia techniques. To the investigators' knowledge no studies since that time have examined FHR monitoring during Cesarean deliveries using external monitoring or spinal anesthesia

ELIGIBILITY:
Inclusion Criteria:

1. First 15 patients only- Elective induction of labor, not yet in active labor.
2. Subsequent 40 patients - Scheduled cesarean sections performed under spinal anesthesia
3. Patients ages 18-45

Exclusion Criteria:

1. Urgent or emergent cesarean sections
2. Cesarean sections performed under general anesthesia

Ages: 18 Years to 45 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Study Population: Pregnant women with scheduled induction of labor and pregnant women with schedule cesarean delivery.
Sampling Method: Non-Probability Sample
Enrollment: 4 (Actual)
Dates: Start 2016-10; Primary Completion 2017-10-29 (Actual); Study Completion 2017-10-29 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Heather McKenzie, MD, Principal Investigator — Washington University School of Medicine
Locations (1):
- Washington University St Louis School of Medicine, St Louis, Missouri, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Intraoperative FHR Monitoring
Started | 4
Completed | 4
Not Completed | 0

BASELINE CHARACTERISTICS:
Population: No results were analyzed.
Arm/Group | Intraoperative FHR Monitoring
Number analyzed (Participants) | 0
Age, Customized
Sex: Female, Male
Race (NIH/OMB)
Region of Enrollment [unit: participants]
external abdomianl wall fetal ECG sensors to assess FHR — The primary endpoint of the feasibility study is the use of external abdominal wall fetal ECG sensors to assess FHR; its use-friendliness, the signal=noise ration and the correleation wtih acoustic data.

OUTCOME MEASURES:

1. Primary Outcome: ECG of Fetal Heart Rate
Description: This measure will be compared to the acoustic monitoring of FHR across the same 10 minutes.
Time Frame: 10 minutes of evaluable ECG reading
Population: The study was terminated and no results were analyzed.
Arm/Group | Intraoperative FHR Monitoring
Number analyzed (Participants) | 0

ADVERSE EVENTS:
Time Frame: Study participation is approximately 1.5 hours.
Arm/Group | Intraoperative FHR Monitoring
All-Cause Mortality (participants affected / at risk) | 0/4
Serious Adverse Events (participants affected / at risk) | 0/4
Other Adverse Events (participants affected / at risk) | 0/4

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2016-10-20): https://cdn.clinicaltrials.gov/large-docs/96/NCT02950896/Prot_SAP_000.pdf
  • Informed Consent Form (2017-06-15): https://cdn.clinicaltrials.gov/large-docs/96/NCT02950896/ICF_001.pdf